CLINICAL TRIAL: NCT01609972
Title: Multi-Center, Prospective, Randomized, Controlled Clinical Trial to Demonstrate Non-Inferiority of the Senza™ Spinal Cord Stimulation (SCS) System in the Treatment of Chronic Pain as Compared to Commercially Available SCS Devices
Brief Title: Comparison of Senza to Commercial Spinal Cord Stimulation for the Treatment of Chronic Pain
Acronym: SENZA-RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nevro Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA2011 US
Record Dates: First submitted 2012-05-30; First posted 2012-06-01 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Low Back Pain
Keywords: Back pain; Spinal Cord Stimulation
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test (Experimental): Subjects randomized to this arm will be trialed and implanted with the Nevro Senza System
  Interventions: Device: Spinal Cord Stimulator
- Control (Active Comparator): Subjects randomized to this arm will be trialed and implanted with a commercially available SCS system.
  Interventions: Device: Spinal Cord Stimulator

INTERVENTIONS:
Device: Spinal Cord Stimulator — Non-inferior comparison of implantable spinal cord stimulators

SUMMARY:
The purpose of this investigational study is to establish the safety and effectiveness of electrical stimulation delivered to the spinal cord in subjects with chronic, intractable pain of the trunk and/or limbs and will be a comparison of the Senza System with commercially available SCS systems.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with chronic, intractable pain of the trunk and/or limbs (VAS ≥ 5) which has been refractory to conservative therapy for a minimum of 3 months.
* Be an appropriate candidate for the surgical procedures required in this study based on the clinical judgment of the implanting physician
* Be 18 years of age or older at the time of enrollment
* Be willing and capable of giving informed consent
* Be willing and able to comply with study-related requirements, procedures, and visits

Exclusion Criteria:

* Have a medical condition or pain in other area(s), not intended to be treated with SCS, that could interfere with study procedures, accurate pain reporting, and/or confound evaluation of study endpoints, as determined by the Investigator
* Have evidence of an active disruptive psychological or psychiatric disorder or other known condition significant enough to impact perception of pain, compliance of intervention and/or ability to evaluate treatment outcome, as determined by a psychologist
* Have a current diagnosis of a coagulation disorder, bleeding diathesis, progressive peripheral vascular disease or uncontrolled diabetes mellitus
* Have a diagnosis of scoliosis that precludes lead placement
* Have an existing drug pump and/or SCS system or another active implantable device such as a pacemaker
* Have prior experience with SCS
* Have a condition currently requiring or likely to require the use of MRI or diathermy
* Have metastatic malignant disease or active local malignant disease
* Have a life expectancy of less than 1 year
* Have an active systemic or local infection
* Be pregnant (if female and sexually active, subject must be using a reliable form of birth control, be surgically sterile or be at least 2 years post-menopausal)
* Have within 6 months of enrollment a significant untreated addiction to dependency producing medications or have been a substance abuser (including alcohol and illicit drugs)
* Be concomitantly participating in another clinical study
* Be involved in an injury claim under current litigation
* Have a pending or approved worker's compensation claim

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2012-06; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Change in back pain VAS and neurological status from Baseline | 3 months
  The primary endpoint is a composite of effectiveness and safety. Specifically, the primary endpoint is the percentage of randomized subjects (the ITT analysis population) and subjects completing the Primary Efficacy Assessment (the PP analysis population) who respond to SCS therapy (as assessed by VAS) for back pain and do not have a stimulation-related neurological deficit at the Primary Efficacy Assessment (non-inferiority analysis). Subjects who do not have a successful Trial Phase are considered failures (non-responders) toward the primary endpoint.

SECONDARY OUTCOMES:
Change in disability as measured by Oswestry Disability Index | 3, 6, 12 months
Number of subjects with adverse events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Kapural, MD, Principal Investigator — The Center for Clinical Research, Winston-Salem, NC

REFERENCES:
- [Derived] Amirdelfan K, Yu C, Doust MW, Gliner BE, Morgan DM, Kapural L, Vallejo R, Sitzman BT, Yearwood TL, Bundschu R, Yang T, Benyamin R, Burgher AH, Brooks ES, Powell AA, Subbaroyan J. Long-term quality of life improvement for chronic intractable back and leg pain patients using spinal cord stimulation: 12-month results from the SENZA-RCT. Qual Life Res. 2018 Aug;27(8):2035-2044. doi: 10.1007/s11136-018-1890-8. Epub 2018 Jun 1. PMID 29858746